CLINICAL TRIAL: NCT04532151
Title: Optical Coherence Tomography Imaging in Systemic Sclerosis
Acronym: OCTISS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 7630
Record Dates: First submitted 2020-07-29; First posted 2020-08-31 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Systemic Sclerosis; Early Systemic Sclerosis Without Clinical Scleroderma and Onset < 2 Years
Keywords: Systemic sclerosis; Scleroderma; Optical coherence tomography (OCT)
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is an open-label study. The mRSS will be performed by an independent clinician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early SSc group (Other): Patients with SSc according to the criteria ACR / EULAR 2013, without scleroderma Normal routine clinical examinations and routine biology tests will be performed. For non-invasive imaging specific to the study, various parameters will be measured on the finger and forearm by LC-OCT, LC-OCT-Doppler, HD ultrasound as well as fluid silicone molding in a dimly lit room. The mRSS will be evaluated by an experienced clinician, blinded from imaging measurements.
  Patients will be reassessed at M24. The participation of each subject will be 24 months, with two visits of one hour.
  The clinical data corresponding to the current practice will be collected in a study specific case report form.
  Interventions: Diagnostic Test: Non-invasive skin imaging assessment
- Established SSc group (Other): Patients with SSc according to criteria ACR / EULAR 2013 with scleroderma Normal routine clinical examinations and routine biology tests will be performed. For non-invasive imaging specific to the study, various parameters will be measured on the finger and forearm by LC-OCT, LC-OCT-Doppler, HD ultrasound as well as fluid silicone molding in a dimly lit room. The mRSS will be evaluated by an experienced clinician, blinded from imaging measurements. The participation of each subject will be one hour.
  The clinical data corresponding to the current practice will be collected in a study specific case report form.
  Interventions: Diagnostic Test: Non-invasive skin imaging assessment
- Control group: (Other): Patient without systemic sclerosis Normal routine clinical examinations and routine biology tests will be performed. For non-invasive imaging specific to the study, various parameters will be measured on the finger and forearm by LC-OCT, LC-OCT-Doppler, HD ultrasound as well as fluid silicone molding in a dimly lit room. The participation of each subject will be one hour.
  The clinical data corresponding to the current practice will be collected in a study specific case report form.
  Interventions: Diagnostic Test: Non-invasive skin imaging assessment

INTERVENTIONS:
Diagnostic Test: Non-invasive skin imaging assessment — Intervention Description : (Limit: 1000 characters) Do not repeat information already included in arm/group descriptions. Specify details not covered in associated Arm
  One session of Non-invasive skin imaging assessment contained:
  * an examination on LC-OCT
  * an examination on LC-OCT-doppler
  * a fluid silicone molding
  * an examination on HD ultrasound
  The measurements will be applied on 3 skin sites: the dorsal surface of the finger, the inner face and the outer surface of the forearm.
  The imaging assessment lasts 30 minutes in a dimly lit room where the humidity and temperature are stable.

SUMMARY:
Systemic sclerosis (SSc) is an autoimmune disorder characterized by early vascular endothelial involvement. SSc is a rare and devastating multi-visceral disease when fibrotic lesions extend to the skin and other tissues (heart, lungs, kidneys). The severity of skin involvement in SSc is correlated with functional prognosis and survival. To date, there is no validated tool for a reliable quantitative assessment of skin fibrosis.

Optical coherence tomography (OCT) is an innovative non-invasive skin imaging technique that allows micrometric analysis of the superficial layers of the skin. Previous study showed that OCT could detect the loss of the dermal-epidermal junction in an objective and non-invasive way, which is correlated with severity of skin fibrosis.

The aim of OCTISS study is to evaluate the skin involvement of patients with early SSc using OCT imaging. This will be early diagnosis of fibrosis lesions and help identify patients at an early stage.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a rare autoimmune disorder. It is characterized by fibrosis and vascular obliteration in the skin and other organs. Skin damage, manifested by thickening of the skin tissue, is often one of the first signs of the disease. Pathogenesis is dominated by early microvascular changes targeting endothelial cells and with the release of several mediators promoting an inflammatory response and vascular remodeling. This inflammatory cascade results in fibrosis lesions. Early diagnosis of fibrosing skin lesions is essential in SSc since their severity is correlated with functional prognosis and survival. To date, there is no validated tool to reliably quantify skin fibrosis. The semi-quantitative Modified Rodnan score (mRSS), based on clinical assessment of skin thickening at 17 anatomical areas, is widely used. The main limitation of this method is its inter-operator variability. The histopathological analysis of the skin biopsy is interesting but invasive. The new non-invasive and reproducible tools are needed to evaluate skin fibrosis for early diagnosis of SSc.

Optical coherence tomography (OCT) is an innovative imaging technique that uses a light wave to capture 3D images of a material that scatters light. OCT allows real-time, direct and high-resolution imaging of the morphology of the biological sample (such as skin) without ionizing radiation. In SSc, the cutaneous fibrosis is characterized by a deregulated production of the components of the extracellular matrix, in particular collagen. Previous results showed that the dermal-epidermal junction could be observed in healthy subjects using OCT. In patients with SSc and skin involvement, the visualization of this junction could be reduced. The results suggest a possible correlation between the intensity of visualization of the dermo-epidermal junction and the severity of cutaneous fibrosis.

In this project, we would like to compare the skin involvement of the dorsal surface of a finger between patients with early SSc and control subjects using non-invasive OCT imaging. The study population meets the criteria for early SCS, with onset of disease less than 2 years and without clinically detectable skin involvement. In a second time, other imaging techniques (HD ultrasound) or fluid silicone molding technique will be used to evaluate the progression of skin fibrosis or the morphological characteristics of the skin or vascular network of the patient with early SSc. To complete the work, these parameters will be evaluated in other anatomical sites (outer and inner side of the forearm) or in another group of patients (Established SSc patients with clinical cutaneous sclerosis) or at another timepoint (M24). The hypothesis of this study is that OCT can be used to identify SSc patients at a stage where the lesions are still early and reversible.

This is a prospective, monocentric, comparative, open-label and longitudinal patient study with duration of 36 months. The duration of the inclusion period will be 12 months. The participation of each subject is from 1 hour (for group 2 and 3) to 24 months (for group 1). We planned to include 60 patients in the Department of Rheumatology of the University Hospital of Strasbourg (20 patients from each group).

The different measures in the study are not invasive. No specific biological sampling of the study will be conducted. There will be no change for the treatment of patients either.

ELIGIBILITY:
IInclusion criteria

* Major subject (age ≥ 18 years)
* Male or female subject
* Subject affiliated to a social health insurance scheme
* Subject having signed an informed consent
* Subject having been informed of the results of the prior medical examination

Inclusion criteria specific to each group

* Group 1 "Early SSc group": Patients with SSc according to ACR / EULAR criteria (2013) early onset <2 years and without clinical cutaneous sclerosis
* Group 2 "Established SSc group": Patients with SSc according to ACR / EULAR criteria (2013) with cutaneous sclerosis
* Group 3 "Control group": Hospitalized patients in the Rheumatology Department of the University Hospitals of Strasbourg, excluding connective tissue disease

Exclusion criteria:

* Non-inclusion criteria for patients / controls in 3 groups
* Subject having undergone a physical treatment (radiotherapy, surgical intervention ...) on the cutaneous sites studied
* Subjects who received general corticosteroid therapy in the last 3 months
* Subjects being treated with topical corticosteroids on the different cutaneous sites studied
* Impossibility to give clear information of subject (subject in emergency situation, subject with difficulties of understanding ...)
* Subject in exclusion period (determined by previous or current study),
* Subject under the protection of justice, guardianship or curatorship
* Pregnancy (on declaration of the patient)

Non-inclusion criteria specific to each group

- Group 1 "Early SSc group": Patients with SSc and having a clinical cutaneous sclerosis

- Group 2 "Established SSc group": Patients with criteria for another systemic autoimmune disease

- Group 3 "Control group":

* Subjects with scleroderma,
* Subjects with Raynaud's phenomenon
* Subjects with other sclerosing disease (morphea, Shulman,…)
* Diabetic subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Optic density of the papillo-reticular dermis on the dorsal surface of a finger | This parameter will be evaluated during a hospital consultation. The test lasts 30 minutes. For all three groups, the measurements will be taken at the time of the inclusion visit (V0)
  The optic density of the papillo-reticular dermis, 300 μm deep, on the dorsal surface of a finger will be measured in all three groups using optical coherence tomography (OCT)
Optic density of the papillo-reticular dermis on the dorsal surface of a finger | Only the patient of group 1 (Early SSc group) will be evaluated again during the visit of Month 24 (V M24).

SECONDARY OUTCOMES:
Optic density of the papillo-reticular dermis at the outer and inner side of the forearm | These parameters will be evaluated during a hospital consultation. The test lasts 30 minutes. For all three groups, the measurements will be taken at the time of the inclusion visit (V0).
  The optic density of the papillo-reticular dermis, 300 μm deep, at the outer and inner side of the forearm will be measured in all three patient groups using OCT.
Optic density of the papillo-reticular dermis at the outer and inner side of the forearm | Only the patient of group 1 (Early SSc group) will be evaluated again during the visit of Month 24 (V M24).
  The optic density of the papillo-reticular dermis, 300 μm deep, at the outer and inner side of the forearm will be measured in all three patient groups using OCT.
Modified Rodnan skin score (mRSS) | The assessment will be applied only to patients in group 1 (Early SSc group) and group 2 (Established SSc group) at the inclusion visit (V0).
  The Modified Rodnan Score (mRSS) will be evaluated by an experienced clinician at each anatomical site studied during a hospital consultation. The test lasts 5 minutes. The evaluator will be blinded from the results of the imaging.
Modified Rodnan skin score (mRSS) | Only the patient of group 1 (Early SSc group) will be evaluated again during the visit of Month 24 (V M24).
The thickness of the hypodermis, obtained by HD ultrasound. | Day 0
The thickness of the dermis, obtained by HD ultrasound | Day 0
The distribution of tension forces exerted within the dermis by fluid silicone molding techniques | Day 0
The optic density of the papillo-reticular dermis, 300 μm deep, at the outer and inner side of the forearm will be measured in all three patient groups using OCT. | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Chatelus, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France